CLINICAL TRIAL: NCT07141576
Title: Comparative Efficacy of Erbium and Diode Laser Systems Alone or Combined With Fluoride-Based Desensitizing Agent in the Management of Dentinal Hypersensitivity: A Randomized Controlled Clinical Trial
Brief Title: Comparative Efficacy of Laser Systems and Fluoride in Managing Dentinal Hypersensitivity: RCT
Acronym: DHLT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayman Mohamed Elamin Taha, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CairoU-Laser Hypersensitivity
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Dentin Sensitivity, Dentine Hypersensitivity, Tooth Sensitivity
Keywords: Sensitivity, Laser, Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity | interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial uses a single-blind, parallel-group design to compare four treatments for dentinal hypersensitivity in 96 participants. Using computer-generated randomization and sealed envelope allocation, participants are equally divided into four groups receiving Erbium laser, Diode laser, combination Diode laser with fluoride, or fluoride alone. The study employs blinded outcome assessors, sham procedures to minimize bias, and follows participants for 6 months with Visual Analogue Scale measurements at baseline, 1 week, 4 weeks, and 6 months to assess treatment effectiveness.
Who Masked: Outcomes Assessor
Masking Description: This randomized controlled trial uses a single-blind, parallel-group design to compare four treatments for dentinal hypersensitivity in 96 participants. Using computer-generated randomization and sealed envelope allocation, participants are equally divided into four groups receiving Erbium laser, Diode laser, combination Diode laser with fluoride, or fluoride alone. The study employs single-blind masking where outcome assessors and statisticians remain blinded to treatment assignments, while sham procedures (simulated laser/fluoride applications) minimize bias where complete blinding is impossible. Participants are followed for 6 months with Visual Analogue Scale measurements at baseline, 1 week, 4 weeks, and 6 months to assess treatment effectiveness using standardized protocols and pre-calibrated examiners.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Erbium Laser (Experimental): Erbium:YAG laser (2940 nm) treatment alone using thermal ablation to seal dentinal tubules and reduce hypersensitivity.
  Interventions: Other: Diode laser (650 nm): Visible red light energy; Drug: Fluoride varnish
- Diode Laser (Experimental): Diode laser (650 nm) photobiomodulation therapy alone targeting neural modulation to reduce pain transmission.
  Interventions: Other: Erbium laser (2940 nm): Infrared light energy; Drug: Fluoride varnish
- Combination Therapy (Experimental): Diode laser (650 nm) followed immediately by fluoride varnish application combining neural modulation with tubule occlusion.
  Interventions: Other: Erbium laser (2940 nm): Infrared light energy; Other: Diode laser (650 nm): Visible red light energy; Drug: Fluoride varnish
- Fluoride Control (Active Comparator): 5% sodium fluoride varnish alone serving as active control, promoting remineralization and tubule occlusion through standard treatment.
  Interventions: Other: Erbium laser (2940 nm): Infrared light energy; Other: Diode laser (650 nm): Visible red light energy

INTERVENTIONS:
Other: Erbium laser (2940 nm): Infrared light energy — The lasers emit light energy in the infrared and visible spectrum, which is fundamentally different from ionizing radiation (like X-rays or gamma rays) that can damage DNA. Dental lasers work through photobiomodulation and thermal effects, not through radiation exposure.
  Arms: Combination Therapy; Diode Laser; Fluoride Control
Other: Diode laser (650 nm): Visible red light energy — Non-ionizing radiation or more accurately as optical energy devices, not ionizing radiation.
  Arms: Combination Therapy; Erbium Laser; Fluoride Control
Drug: Fluoride varnish — Biological Intervention
  Arms: Combination Therapy; Diode Laser; Erbium Laser

SUMMARY:
This randomized controlled clinical trial aims to compare the effectiveness of Erbium laser (2940 nm), Diode laser (650 nm), combination Diode laser with fluoride varnish, and fluoride varnish alone in treating dentinal hypersensitivity. The study will recruit 96 adults aged 18-45 years with tooth sensitivity scores ≥4 on a 0-10 Visual Analogue Scale, randomly allocating 24 participants to each of four treatment groups. The primary outcome is reduction in tooth sensitivity measured at baseline, 1 week, 4 weeks, and 6 months post-treatment, with patient satisfaction as a secondary outcome. Conducted at Cairo University's Faculty of Dentistry, this 6-month follow-up study addresses the limitation of current treatments that provide only temporary relief, seeking to establish evidence-based protocols for optimal long-term management of dentinal hypersensitivity by evaluating whether laser therapies alone or in combination with fluoride offer superior and more durable pain relief compared to standard fluoride treatment alone.

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigates the comparative efficacy of different laser systems and fluoride-based treatments for managing dentinal hypersensitivity, a prevalent clinical condition characterized by sharp, transient pain from exposed dentin in response to thermal, evaporative, tactile, or chemical stimuli. The study will recruit 96 participants aged 18-45 years with dentinal hypersensitivity scores ≥4 on a Visual Analogue Scale (VAS), randomly allocating them into four equal groups (n=24 each): Group 1 receiving Erbium:YAG laser treatment (2940 nm, 80mJ, 2Hz) which works through thermal tubule occlusion; Group 2 receiving Diode laser photobiomodulation therapy (650 nm, 100mW, 2J total dose) targeting neural modulation; Group 3 receiving combination therapy of Diode laser with 5% sodium fluoride varnish to exploit synergistic mechanisms; and Group 4 receiving fluoride varnish alone as the control comparator. The primary outcome measures dentinal hypersensitivity reduction using VAS scores (0-10 scale) assessed through standardized evaporative stimulus tests at baseline, 1 week, 4 weeks, and 6 months post-treatment, while secondary outcomes include patient satisfaction and treatment tolerability. Conducted at the Conservative Dentistry Department, Faculty of Dentistry, Cairo University, with blinded outcome assessors and standardized protocols, this superiority trial addresses the clinical need for evidence-based, long-term effective treatments for dentinal hypersensitivity by comparing individual laser modalities against combination therapy and established fluoride treatments, potentially establishing optimal therapeutic protocols that provide both immediate relief and sustained tubule occlusion or neural modulation for improved patient quality of life.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18-45 years
* Both sexes eligible
* Good general health status
* At least one tooth with cervical dentin hypersensitivity (CDH)
* Visual Analogue Scale (VAS) pain score ≥ 4 on evaporative stimulus test using dental syringe air jet
* Willing to participate and provide informed consent

Exclusion Criteria

* Active carious lesions or defective restorations requiring treatment
* Loss of dental tissue requiring restorative treatment
* Previous professional desensitizing treatment within 6 months prior to recruitment
* Use of desensitizing toothpastes within 3 months prior to study
* Current use of anti-inflammatory drugs or analgesics at time of recruitment
* Pregnant or breastfeeding women
* Inability to comply with study protocol or follow-up requirements

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Dentinal Hypersensitivity Assessment | at baseline, 1 week, 4 weeks, and 6 months post-treatment
  Dentinal Hypersensitivity Assessment Using Visual Analogue Scale

SECONDARY OUTCOMES:
Patient Satisfaction | at baseline, 1 week, 4 weeks, and 6 months post-treatment
  The secondary outcome measures patient satisfaction with treatment using a categorical Yes/No assessment. Participants report their overall satisfaction with the assigned intervention based on perceived pain relief.

IPD SHARING:
Plan to Share IPD: No